CLINICAL TRIAL: NCT04074148
Title: Effectiveness of Diabetes Prevention Education Program on Diabetes Prevention Among Prediabetes Population in Nepal: A Cluster Randomized Controlled Trial
Brief Title: Effectiveness of Diabetes Prevention Education Program on Diabetes Prevention Among Prediabetes Population in Nepal
Acronym: DiPEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/783
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Prediabetic State
Keywords: Patient Education; Nepal; Diabetes prevention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Education Program (Experimental): Diabetes Prevention Education Program
  Interventions: Behavioral: Diabetes Prevention Education Program
- control (Experimental): Diabetes Prevention Education brochure
  Interventions: Behavioral: Diabetes Prevention Education brochure

INTERVENTIONS:
Behavioral: Diabetes Prevention Education Program — An educational lifestyle modification program, offering 4 sessions of 30 minutes theory and 30 minutes practice each, total duration 6 months
  Arms: Diabetes Prevention Education Program
Behavioral: Diabetes Prevention Education brochure — An educational lifestyle modification brochure
  Arms: control

SUMMARY:
Background: The prediabetes population is a high risk group for developing diabetes and is also associated with a higher risk of micro- and macrovascular complications. Prevalence of prediabetes is also increasing in Nepal (10.3%). Therefore, appropriate strategies should be developed to detect prediabetes and prevent its complications. Early detection of prediabetes offers opportunity for intervention to prevent diabetes either by reverting into normoglycemia or stabilizing blood glucose levels. Even a small shift in weight loss and reduction of glycated haemoglobin (HbA1c) (i.e., a change in HbA1c of 0.5%) can be significant in reducing cardiometabolic risk. Therefore, we propose to develop a culturally tailored Diabetes Prevention Education Program (DiPEP) for Nepal and implement this program among a prediabetes population with the aim to prevent diabetes.

Aims: Primary aim of the research is to test the effectiveness of a Diabetes Prevention Education Program (DiPEP) in lowering glycated haemoglobin (HbA1c %) among a pre-diabetes population in Nepal. Our secondary aims are to test the effectiveness of DiPEP in improving health literacy in diabetes, reducing weight, improving healthy diet and physical activity. We also aim to explore acceptability and usability of DiPEP among a prediabetes population and perception of adoption and sustainability of DiPEP in the health sector of Nepal.

Significance: Prevention of diabetes, especially Type 2 Diabetes Mellitus (T2DM) is proven, possible and powerful. It is more cost effective than spending huge money in treatment and usual care. It requires modification of dietary and exercise behavior, which are efficacious, safe, and cost-effective measures. Therefore, a culturally tailored DiPEP intervention program for Nepal will serve as an additional reference resource for the Non-Communicable Disease division of Ministry of health to develop and implement national diabetes prevention program if they decide such program is important for Nepal. It will be helpful to achieve Non-communicable disease target 3.4 of the Sustainable Development Goal by Nepal government's Ministry of Health. Additionally, it will be beneficial for the prediabetes population who could have developed T2DM in short span of time if they had been undiagnosed and unconsidered. Therefore, the main significance of the study is it will provide knowledge and environment to prevent diabetes at their community level.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents of Dhulikhel municipality or Lalitpur Metropolitan City (Patan)
* Indian Diabetes Risk Score 60 or higher
* Prediabetes: glycated haemoglobin (HbA1c) 5.7-6.4 %
* Random blood sugar ≥ 140 to ≤ 250 mg/dl

Exclusion Criteria:

* type 1 diabetes (self-report)
* Type 2 diabetes
* Under medication
* HbA1c criteria (≥ 6.5 %)
* Currently pregnant
* Critically ill patients

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 291 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
glycated haemoglobin (HbA1c) percent | 6 months
  testing capillary blood sugar by point of care HbA1c Analyser

CONTACTS AND LOCATIONS:
Overall Officials: Bård E Kulseng, phd prof, Study Director — Norwegian University of Science and Technology NTNU
Locations (1):
- Kathmandu University School of Medical Science, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shakya P, Shrestha A, Bajracharya M, Shrestha A, Kulseng BE, Karmacharya BM, Shrestha S, Das S, Shrestha IB, Barun K, Shrestha N, Skovlund E, Sen A. Effectiveness of a group-based Diabetes Prevention Education Program (DiPEP) in a population with pre-diabetes: a cluster randomised controlled trial in Nepal. BMJ Nutr Prev Health. 2023 Dec;6(2):253-263. doi: 10.1136/bmjnph-2023-000702. Epub 2023 Nov 7. PMID 38264365
- [Derived] Shakya P, Shrestha A, Karmacharya BM, Shrestha A, Kulseng BE, Skovlund E, Sen A. Prevalence of prediabetes and associated factors of prediabetic stages: a cross-sectional study among adults in Nepal. BMJ Open. 2022 Dec 29;12(12):e064516. doi: 10.1136/bmjopen-2022-064516. PMID 36581426
- [Derived] Shakya P, Shrestha A, Karmacharya BM, Shrestha A, Kulseng BE, Skovlund E, Sen A. Diabetes Prevention Education Program in a population with pre-diabetes in Nepal: a study protocol of a cluster randomised controlled trial (DiPEP). BMJ Open. 2021 Nov 24;11(11):e047067. doi: 10.1136/bmjopen-2020-047067. PMID 34819277